CLINICAL TRIAL: NCT06155786
Title: Cognitive Effects of Transcranial Direct Current Stimulation (tDCS) and Transcranial Random Noise Stimulation (tRNS) in Schizophrenia: A Random, Crossover Study
Brief Title: Cognitive Effects of tDCS and tRNS in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The National Brain Mapping Laboratory (NBML) (Other)
Collaborators: Leibniz Research Centre for Working Environment and Human Factors (Other); Payame Noor University (Unknown)
Responsible Party: Principal Investigator, Mohammad Ali Salehinejad, Principal Investigator, The National Brain Mapping Laboratory (NBML)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ifado-PNU
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia; Cognitive Impairment
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS group (Active Comparator): In tDCS, direct electrical currents at the intensity of 2 mA are generated by an electrical stimulator and are noninvasively delivered to the left and right dorsolateral prefrontal cortex through a pair of saline-soaked sponge electrodes (7×5 cm) for 30 minutes.
  Interventions: Device: transcranial direct current stimulation (tDCS) active stimulator
- tRNS group (Active Comparator): In tRNS, direct electrical currents at the intensity of 2 mA amplitude (offset at 1 mA) and frequency of 100-640 Hz are generated by an electrical stimulator and are noninvasively delivered to the left and right dorsolateral prefrontal cortex through a pair of saline-soaked sponge electrodes (7×5 cm) for 30 minutes.
  Interventions: Device: transcranial random noise stimulation (tRNS)
- sham group (Sham Comparator): In sham group, placebo stimulation is generated by an electrical stimulator and is noninvasively delivered to the left and right dorsolateral prefrontal cortex through a pair of saline-soaked sponge electrodes (7×5 cm) for 30 minutes.
  Interventions: Device: transcranial direct current stimulation (tDCS) sham stimulator

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) active stimulator — In tDCS the electrical current is applied directly between electrodes mounted on the head which can can de-or hyperpolarizes resting membrane potential and thereby modulate cortical excitability
  Arms: tDCS group
Device: transcranial random noise stimulation (tRNS) — Here, an alternating electrical current is applied at a mix of frequencies it is called transcranial random noise stimulation (tRNS), which can be delivered in low (between 0.1-100 Hz) or high (between 101-640 Hz) frequency stimulation
  Arms: tRNS group
Device: transcranial direct current stimulation (tDCS) sham stimulator — Here a sham electrical current is applied directly between electrodes mounted on the head which can can de-or hyperpolarizes resting membrane potential and thereby modulate cortical excitability
  Arms: sham group

SUMMARY:
The purpose of this study is to investigate the cognitive effects of different electrical stimulation modalities, such as transcranial direct and random-noise stimulation over the dorsolateral prefrontal cortex, in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia based on Diagnostic and Statistical Manual (DSM)5
* Being 18-50 years old (male and female)
* If female, negative urine pregnancy test
* feasibility for tDCS/tRNS interventions according to safety guidelines
* stable medication regime, especially for classical neuroleptics and all central nervous system activating medications, if taken, 4-6 weeks before the experiment
* fluency in the native language
* right-handed
* Required written informed consent signed by patients' guardian

Exclusion Criteria:

* pregnancy
* alcohol or substance dependence
* comorbid bipolar disorder and mood disorder
* history of seizure
* history of neurological disorder
* history of head injury
* Presence of ferromagnetic objects in the body that are contraindicated for brain stimulation of the head (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Spatial Working Memory behavioral performance | During procedure (4 minutes)
  The test begins with a number of coloured squares (boxes) shown on the screen. The aim of this test is that by selecting the boxes and using a process of elimination, the participant should find one yellow 'token' in each of a number of boxes and use them to fill up an empty column on the right-hand side of the screen.
executive function behavioral performance | During procedure (8-10 minutes)
  The participant is shown two displays containing three coloured balls. The test administrator first demonstrates to the participant how to move the balls in the lower display to copy the pattern in the upper display and completes one demonstration problem, where the solution requires one move. The participant must then complete three further problems, one each requiring two moves, three moves, and four moves. Next, the participant is shown further problems and must work out in their head how many moves the solutions require and then select the appropriate box at the bottom of the screen to indicate their response
The Positive and Negative Affect Schedule (PANAS) | through study completion, an average of 3 weeks
  The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire that consists of two 10-item scales to measure both positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much).

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Payame Noor University, Tehran Branch, Tehran
  - Zanjan University, Zanjān

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jafari E, Moghadamzadeh A, Vaziri Z, Atadokht A, Fathi Jouzdani A, Cohen Kadosh R, Nitsche MA, Blumberger DM, Salehinejad MA. Cognitive and emotional effects of bilateral prefrontal anodal tDCS and high-frequency tRNS in schizophrenia: a randomized sham-controlled study. Schizophrenia (Heidelb). 2026 Jan 13. doi: 10.1038/s41537-025-00720-z. Online ahead of print. PMID 41530140